CLINICAL TRIAL: NCT00005810
Title: A Phase II Study of Estramustine, Docetaxel, and Carboplatin With G-CSF Support in Men With Hormone Refractory Prostate Cancer
Brief Title: Combination Chemotherapy Plus Filgrastim in Treating Patients With Stage IV Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-99813; U10CA031946 (NIH); CDR0000067811 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-06-02; First posted 2004-04-19 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Filgrastim; Carboplatin; Docetaxel; Estramustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Estramustine + docetaxel + carboplatin+ filgrastim (Experimental): Patients receive oral estramustine 3 times daily on days 1-5. Patients receive docetaxel IV over 1 hour followed by carboplatin IV over 1 hour on day 2. Filgrastim (G-CSF) SC is administered beginning on day 6 and continuing until hematopoietic recovery. Treatment continues every 21 days in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for a maximum of 2 years.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: docetaxel; Drug: estramustine phosphate sodium

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: docetaxel
Drug: estramustine phosphate sodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus filgrastim in treating patients who have stage IV prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate (objective and PSA response) and duration of response to estramustine, docetaxel, and carboplatin with filgrastim (G-CSF) support in patients with hormone refractory prostate cancer. II. Determine the toxicity of this regimen in this patient population.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IV adenocarcinoma of the prostate Failure on standard hormone therapy Measurable disease with any PSA Accurately measured in at least 1 dimension as at least 20 mm by physical exam for clinically palpable lymph nodes and superficial skin lesions or chest x-ray for clearly defined lung lesions surrounded by aerated lung OR those lesions measured as at least 10 mm by spiral CT scan OR Nonmeasurable disease with PSA at least 5 ng/mL Nontarget lesions including small lesions with longest diameter less than 20 mm by conventional techniques or less than 10 mm by spiral CT scan and truly nonmeasurable lesions including: Bone lesions Pleural or pericardial effusions Ascites CNS lesions Leptomeningeal disease Irradiated lesions unless progression documented after radiotherapy Documented progressive systemic disease despite at least 1 endocrine manipulation with either orchiectomy or LHRH agonist (which must be continued), or diethylstilbestrol For measurable disease: Objective evidence of increase of greater than 20% in the sum of the longest diameters of target lesions from the time of maximal regression or the appearance of 1 or more new lesions For nonmeasurable disease: If bone only disease, appearance of 1 new lesion on bone scan attributable to prostate cancer along with a PSA of at least 5 ng/mL OR An elevated PSA (at least 5 ng/mL) that has risen serially from baseline on 2 occasions each at least 1 week apart Testosterone no greater than 50 ng/mL if no prior bilateral orchiectomy

PATIENT CHARACTERISTICS: Age: 18 to 99 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.0 times upper limit of normal (ULN) AST no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No myocardial infarction or significant change in anginal pattern within past 1 year No congestive heart failure No New York Heart Association class II-IV heart disease No deep venous thrombosis or pulmonary embolus within past 1 year Other: Fertile patients must use effective contraception No clinically significant peripheral neuropathy No known hypersensitivity to E. coli derived products

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent sargramostim (GM-CSF) Chemotherapy: No prior chemotherapy No prior estramustine or suramin No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 4 weeks since prior antiandrogens Primary testicular androgen suppression (e.g., with an LHRH analogue) should not be discontinued Concurrent LHRH analogue allowed if no prior bilateral orchiectomy Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiation and recovered At least 8 weeks since prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium No concurrent palliative radiotherapy Surgery: See Disease Characteristics At least 4 weeks since prior major surgery and recovered

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-03; Primary Completion 2003-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Oh, MD, Study Chair — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina

REFERENCES:
- [Result] Oh WK, Halabi S, Kelly WK, Werner C, Godley PA, Vogelzang NJ, Small EJ; Cancer and Leukemia Group B 99813. A phase II study of estramustine, docetaxel, and carboplatin with granulocyte-colony-stimulating factor support in patients with hormone-refractory prostate carcinoma: Cancer and Leukemia Group B 99813. Cancer. 2003 Dec 15;98(12):2592-8. doi: 10.1002/cncr.11829. PMID 14669278
- [Result] Oh WK, Halabi S, Kelly WK, et al.: A phase II study of estramustine, docetaxel, and carboplatin (EDC) with G-CSF support in men with hormone refractory prostate cancer (HRPC): CALGB 99813. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-779, 2002.